CLINICAL TRIAL: NCT06973005
Title: An Open-label, Fixed Sequence Study in Healthy Participants to Assess the Effect of Multiple Doses of AZD2389 on the Pharmacokinetics of Midazolam, Caffeine, and Bupropion
Brief Title: A Study to Investigate How Multiple Oral Doses of AZD2389 Affect the Pharmacokinetics of Midazolam, Caffeine, and Bupropion in Healthy Participants
Acronym: CRIOLLO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7930C00007
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Advanced Chronic Liver Disease; Healthy Participants
Keywords: Hepatic Fibrosis; FAP inhibitor
MeSH Terms: conditions — Liver Cirrhosis | interventions — Midazolam; Caffeine; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): In Period 1, participants will receive midazolam and caffeine in combination on Day 1. Participants will receive bupropion on Day 2.
  In Period 2, participants will receive AZD2389 for 9 days from Day 5 to Day 13. In Period 3, participants will first receive AZD2389 with midazolam and caffeine in combination on Day 14. On Day 15, participants will first receive AZD2389 with bupropion. On Days 16 and 17, participants will receive AZD2389.
  Interventions: Drug: AZD2389; Drug: Midazolam; Drug: Caffeine; Drug: Bupropion

INTERVENTIONS:
Drug: AZD2389 — Oral dose on Days 5 to 13, Day 16, and Day 17. On Day 14 co-administered with a combination of midazolam and caffeine. On Day 15 co-administered with bupropion.
Drug: Midazolam — Single oral dose on:
  * Day 1 (co-administered with caffeine)
  * Day 14 (co-administered with caffeine and AZD2389)
Drug: Caffeine — Single oral dose on:
  * Day 1 (co-administered with midazolam)
  * Day 14 (co-administered with midazolam and AZD2389)
Drug: Bupropion — Single oral dose on:
  * Day 2 (alone)
  * Day 15 (co-administered with AZD2389)

SUMMARY:
The purpose of this study is to measure the effect of multiple doses of AZD2389 on the pharmacokinetics (PK) of midazolam, caffeine, and bupropion in healthy participants.

DETAILED DESCRIPTION:
This study is an open-label, fixed sequence, 3-period, drug-drug interaction (DDI) study in healthy participants performed at a single Clinical Unit.

The study will comprise:

* A Screening Period of maximum 28 days.
* A Treatment Phase, separated into 3 different periods. Period 1 (Day -2 to Day 4): Participants will receive midazolam and caffeine in combination on Day 1. Participants will receive bupropion on Day 2.

Period 2 (Day 5 to Day 13): Participants will receive AZD2389 for 9 days. Period 3 (Day 14 to Day 18): Participants will first receive AZD2389 with midazolam and caffeine in combination on Day 14. On Day 15, participants will first receive AZD2389 with bupropion. On Days 16 and 17, participants will receive AZD2389.

- A final Follow-up Visit, 7 to 14 days after the last AZD2389 PK sample is taken in Period 3.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Participants with suitable veins for cannulation or repeated venipuncture.
* Have a body mass index (BMI) between 18 and 32 kilograms per meter squared (kg/m2) inclusive and weigh at least 50 kilograms (kg) at Screening.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Any clinically important abnormalities in clinical chemistry, coagulation, hematology, or urinalysis results.
* Any positive result at the Screening Visit for serum hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
* Abnormal vital signs, after 10 minutes supine rest, at the Screening Visit and/or admission to the Clinical Unit (Day -2).
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead safety ECG.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* History of hypersensitivity to DPP4 inhibitors, as judged by the investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to DPP4 inhibitors.
* History of severe dermatological disorders, eg, bullous pemphigoid or Stevens-Johnson syndrome, as judged by the investigator.
* Participants who have previously received AZD2389 within the last 12 months prior to the Screening Visit.
* Known hypersensitivity or previous adverse events associated with midazolam, caffeine, or bupropion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Ratio of treatment to reference based on Cmax (RCmax) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To assess the PK parameter RCmax for midazolam, caffeine, and bupropion in combination with AZD2389 compared to midazolam, caffeine, and bupropion alone.
Ratio of treatment to reference based on AUCinf (RAUCinf) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To assess the PK parameter RAUCinf for midazolam, caffeine, and bupropion in combination with AZD2389 compared to midazolam, caffeine, and bupropion alone.
Ratio of treatment to reference based on AUClast (RAUClast) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To assess the PK parameter RAUClast for midazolam, caffeine, and bupropion in combination with AZD2389 compared to midazolam, caffeine, and bupropion alone.
Ratio of area under concentration-curve from time 0 to 24 hours post-dose (AUC0-24) | Period 1: Days 1-3; Period 3: Days 15-18.
  To assess the PK parameter ratio of AUC0-24 for caffeine in combination with AZD2389 compared to caffeine alone.

SECONDARY OUTCOMES:
Apparent total body clearance (CL/F) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To describe the plasma PK of midazolam, caffeine, bupropion, and their metabolites (1'-OH-midazolam, paraxanthine, and hydroxy-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389. To describe the plasma PK of AZD2389 after multiple dose administration.
Apparent volume of distribution based on the terminal phase (Vz/F) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To describe the plasma PK of midazolam, caffeine, bupropion, and their metabolites (1'-OH-midazolam, paraxanthine, and hydroxy-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389. To describe the plasma PK of AZD2389 after multiple dose administration.
Terminal elimination half-life (t1/2λz) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To describe the plasma PK of midazolam, caffeine, bupropion, and their metabolites (1'-OH-midazolam, paraxanthine, and hydroxy-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389. To describe the plasma PK of AZD2389 after multiple dose administration.
Terminal rate constant (λz) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To describe the plasma PK of midazolam, caffeine, bupropion, and their metabolites (1'-OH-midazolam, paraxanthine, and hydroxy-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389. To describe the plasma PK of AZD2389 after multiple dose administration.
Time to reach maximum observed concentration (tmax) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To describe the plasma PK of midazolam, caffeine, bupropion, and their metabolites (1'-OH-midazolam, paraxanthine, and hydroxy-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389. To describe the plasma PK of AZD2389 after multiple dose administration.
Maximum observed concentration (Cmax) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To describe the plasma PK of midazolam, caffeine, bupropion, and their metabolites (1'-OH-midazolam, paraxanthine, and hydroxy-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389. To describe the plasma PK of AZD2389 after multiple dose administration.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To describe the plasma PK of midazolam, caffeine, bupropion, and their metabolites (1'-OH-midazolam, paraxanthine, and hydroxy-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389. To describe the plasma PK of AZD2389 after multiple dose administration.
Area under concentration-time curve from time 0 to infinity (AUCinf) | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To describe the plasma PK of midazolam, caffeine, bupropion, and their metabolites (1'-OH-midazolam, paraxanthine, and hydroxy-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389. To describe the plasma PK of AZD2389 after multiple dose administration.
AUC0-24 | Period 1: Days 1-3; Period 3: Days 15-18.
  To describe the plasma PK of caffeine and its metabolites (paraxanthine) when caffeine is administered alone and in combination with AZD2389.
RCmax | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To assess the RCmax for the metabolites of midazolam, caffeine, and bupropion (1'-OH-midazolam, paraxanthine, OH-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389.
RAUCinf | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To assess the RAUCinf for the metabolites of midazolam, caffeine, and bupropion (1'-OH-midazolam, paraxanthine, OH-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389.
RAUClast | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To assess the RAUClast for the metabolites of midazolam, caffeine, and bupropion (1'-OH-midazolam, paraxanthine, OH-bupropion) when midazolam, caffeine, or bupropion is administered alone and in combination with AZD2389.
Ratio of treatment to reference based on AUC0-24 (RAUC0-24) | Period 1: Days 1-3; Period 3: Days 15-18.
  To assess the RAUC0-24 for the metabolites of caffeine, (paraxanthine) when caffeine is administered alone and in combination with AZD2389.
Metabolite to parent ratio of the AUCinf | Period 1: Days 1-4; Period 2: Days 5-13; Period 3: Days 14-18.
  To assess the metabolite to parent ratio of the AUCinf for midazolam, caffeine, and bupropion.
Metabolite to parent ratio of the AUC0-24 | Period 1: Days 1-3; Period 3: Days 15-18.
  To assess the metabolite to parent ratio of the AUC0-24 for caffeine and its metabolite (paraxanthine) when caffeine is administered alone and in combination with AZD2389.
Area under concentration-time curve in the dose interval (AUCtau) | Period 2: Days 5-13; Period 3: Day 14.
  To describe the plasma PK of AZD2389 after multiple dose administration.
Observed lowest concentration before the next dose is administered (Ctrough) | Period 2: Days 5-13; Period 3: Day 14.
  To describe the plasma PK of AZD2389 after multiple dose administration.
Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Only SAE: -30 to -3 to Day -1. AE and SAE: From Day 1 to Follow-up/Early Termination Visit (Days 25-32)
  To assess the safety and tolerability of multiple oral doses of AZD2389 alone or in combination with midazolam, caffeine and bupropion in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/